CLINICAL TRIAL: NCT00574301
Title: Percutaneous Removal and Margin Ablation for Breast Cancer
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of Arkansas (Other)
Collaborators: Department of Health and Human Services (U.S. Federal Agency); Ethicon Endo-Surgery (Industry); RITA Medical Systems (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UAMS 07050; NIH Grant 5 R21 CA097715-01
Record Dates: First submitted 2007-12-14; First posted 2007-12-17 (Estimated); Last update posted 2013-07-25 (Estimated); Status verified 2013-07

CONDITIONS: Breast Cancer
Keywords: Image Guided Vacuum Assisted Biopsy; Radiofrequency Ablation; Breast Conservation Therapy; Mastectomy; MRI
MeSH Terms: conditions — Breast Neoplasms | interventions — Radiofrequency Ablation; Mastectomy, Segmental; Mastectomy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental)
  Interventions: Procedure: Percutaneous Removal and Margin Ablation

INTERVENTIONS:
Procedure: Percutaneous Removal and Margin Ablation — Patients with a diagnosis of unicentric invasive breast cancer diagnosed by IVEB will then be assigned to the next available surgery date. On that day, the patient's axillary staging will be done, followed by ablation of the biopsy cavity using RFA. The breast surgery may include lumpectomy (which will be directed with US-guidance to assure more accurate removal of the en bloc IVEB site and the margin zone of ablation) or simple mastectomy with or without reconstruction. The tissue specimen will be sent immediately from the operating room to Pathology for routine processing.
  Other Names: Mammotome Breast Biopsy System (IVEB), Ethicon Endo-Surgery; Radiofrequency Ablation (RFA), RITA Medical Systems; Lumpectomy; Mastectomy

SUMMARY:
We hypothesize that radiofrequency ablation after single-insertion image guided vacuum assisted biopsy (IVEB) can be used to achieve negative margins in small unicentric breast cancers (≤1.5 cm).

DETAILED DESCRIPTION:
Using the Mammotome Breast Biopsy System (IVEB) in conjunction with MRI to predict extent of disease, ultrasound to direct removal of the tumor, touch preparation cytology for diagnosis, and ablation of margins using radiofrequency ablation (RFA), we propose to develop a comprehensive system for same-day diagnosis and treatment of patients with small breast lesions.

ELIGIBILITY:
Inclusion Criteria:

* Female, 18 to 90 years of age
* Non-pregnant, not breastfeeding
* Pre-study documentation of:
* Size ≤1.5 cm cancer successfully removed by US-guided IVEB within 30 days of registration
* Uni-centricity, unilateral cancer by radiology (mammogram and MRI)
* Location of abnormality > 1 cm from the skin
* Ductal Carcinoma, Invasive (Grade I-III) or In-Situ
* No palpable axillary or supraclavicular lymph nodes
* Good general health
* Zubrod Performance Status of 0, 1, or 2
* If prior non-breast malignancy, must have 5 year disease-free survival
* No prior chemotherapy
* Hormonal therapy must be stopped
* Therapy with tamoxifen must have been of 14 days or less duration

Exclusion Criteria:

* Subjects less than 18 years of age or greater than 90 years of age
* Pregnant or breastfeeding
* Male
* Prior Breast Biopsy affected breast
* Breast implants
* Multicentric disease, bilateral disease
* Residual disease after IVEB of > 1cm on MRI
* Lesions > 1.5 cm in diameter
* Lesions < 1 cm from skin surface
* Previous radiation therapy to the breast

Ages: 18 Years to 90 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2002-03; Primary Completion 2007-10 (Actual); Study Completion 2011-10 (Actual)

PRIMARY OUTCOMES:
To quantify the degree of tumor-free margin achieved with image-guided vacuum assisted biopsy followed by ablation with radiofrequency ablation | Post-surgical pathology review

SECONDARY OUTCOMES:
The proportion of patients with viable tumor cells beyond the margin | Post-surgical pathology review

CONTACTS AND LOCATIONS:
Overall Officials: V. Suzanne Klimberg, MD, Principal Investigator — University of Arkansas
Locations (1):
- University of Arkansas For Medical Sciences, Little Rock, Arkansas, United States

REFERENCES:
- [Background] Johnson AT, Henry-Tillman RS, Smith LF, Harshfield D, Korourian S, Brown H, Lane S, Colvert M, Klimberg VS. Percutaneous excisional breast biopsy. Am J Surg. 2002 Dec;184(6):550-4; discussion 554. doi: 10.1016/s0002-9610(02)01099-1. PMID 12488164
- [Result] Klimberg VS, Boneti C, Adkins LL, Smith M, Siegel E, Zharov V, Ferguson S, Henry-Tillman R, Badgwell B, Korourian S. Feasibility of percutaneous excision followed by ablation for local control in breast cancer. Ann Surg Oncol. 2011 Oct;18(11):3079-87. doi: 10.1245/s10434-011-2002-y. Epub 2011 Sep 9. PMID 21904959